CLINICAL TRIAL: NCT04200235
Title: Study on Pharmacokinetics and Clinical Efficacy of Dexmedetomidine Hydrochloride Nasal Spray for Preoperative Sedation in Children
Brief Title: A Trial of Dexmedetomidine Hydrochloride Nasal Spray in Preoperative Sedation of Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR0171401-102
Record Dates: First submitted 2019-11-25; First posted 2019-12-16 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2019-11

CONDITIONS: Preoperative Sedation

STUDY DESIGN:
Intervention Model Description: Dexmedetomidine hydrochloride nasal spray compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High weight group (Experimental): High weight group
  Interventions: Drug: Dexmedetomidine hydrochloride nasal spray; Drug: Dexmedetomidine hydrochloride nasal spray blank preparation.
- Low weight group (Experimental): Low weight group
  Interventions: Drug: Dexmedetomidine hydrochloride nasal spray; Drug: Dexmedetomidine hydrochloride nasal spray blank preparation.

INTERVENTIONS:
Drug: Dexmedetomidine hydrochloride nasal spray — In the low weight group, 18 subjects will receive a low dose of dexmedetomidine nasal spray.
  In the high weight group, 18 subjects will receive a high dose of dexmedetomidine nasal spray.
Drug: Dexmedetomidine hydrochloride nasal spray blank preparation. — In the low weight group, 6 subjects will receive dexmedetomidine hydrochloride nasal spray blank preparation.
  In the high weight group, 6 subjects will receive dexmedetomidine hydrochloride nasal spray blank preparation.
  Other Names: Placebo

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and the population pharmacokinetic characteristics of dexmedetomidine hydrochloride nasal spray for preoperative sedation in children

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Male or female
3. Subjects requiring elective general anesthesia surgery
4. Conform to the ASA Physical Status Classification
5. Meet the weight standard

Exclusion Criteria:

1. Not suitable for nasal spray
2. Pediatric populations requiring special care or court/social welfare supervision
3. Subjects who had been under general anesthesia were randomized
4. Subjects with mental disorders and cognitive impairment；Subject with a history of epilepsy
5. Subjects with previous abnormal behavior after medication
6. Subjects with cardiovascular disease
7. Clinically significant abnormal clinical laboratory test value
8. Subjects whose hemoglobin is below the lower limit of normal
9. Subjects who have either an adrenergic receptor agonist or an antagonist were randomized
10. Participated in clinical trials of other drugs before screening (accepted experimental drugs)
11. A history or possibility of difficult airway
12. History of hypersensitivity to drug ingredients or components
13. Other circumstances that the investigator judged inappropriate for participation in this clinical trial

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
PK Cmax | 0 to 1 hour after administration
  Maximum blood concentration (Cmax)

SECONDARY OUTCOMES:
Proportion of subjects who parent-child separation successful | 0 minute to 45 minutes after administration: every 15 minutes after administration
  The FUNK scale is a scale of 1 to 4 for sedation, anxiety, and separation from parents. Separation success defined as a scale of 3 or 4 per item.
Proportion of subjects who the Ramsay score is satisfactory at least once | 0 minute to 45 minutes after administration: every 5 minutes after administration
  Sedation level using the Ramsay scale. Ramsay Satisfaction defined as a scale of 2, 3, or 4;
Proportion of subjects who the UMSS Scale is satisfactory at least once | 0 minute to 45 minutes after administration: every 5 minutes after administration
  Sedation level using the University of Michigan Sedation Scale. UMSS satisfaction defined as a scale of 3, 4, 5, or 6;
Total consumption of propofol(mg) during general anesthesia | From the beginning of anesthesia to the end of surgical operation up to 4 hours
  Total consumption of propofol(mg) during general anesthesia
Total consumption of opioid analgesic(μg) during general anesthesia | From the beginning of anesthesia to the end of surgical operation up to 4 hours
  Total consumption of opioid analgesic(μg) during general anesthesia
Time of anesthesia awakening | Up to 4 hours after the end of surgical operation
  Time of anesthesia awakening
Proportion of subjects with postoperative agitation | Up to 4 hours after the end of surgical operation
  Proportion of subjects with postoperative agitation

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing children's hospital, capital medical university, Beijing, Beijing Municipality, China